CLINICAL TRIAL: NCT02686333
Title: Meditation Intervention for the Treatment of Depression and Anxiety Symptoms in Patients Undergoing Dialysis: A Randomized Control Trial
Brief Title: Meditation for Depression and Anxiety Symptoms in Dialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Collaborators: University Health Network, Toronto (Other); Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Karl Looper, MD, FRCPC, Chief of the Department of Psychiatry, Jewish General Hospital, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-160
Record Dates: First submitted 2015-12-30; First posted 2016-02-19 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Depression; Anxiety
Keywords: Meditation; Dialysis
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Meditation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Meditation Intervention Arm (Experimental): 10-15 minute meditation practices (brief silent meditations, guided meditations, body scans, gentle arm movement exercises). Before each session, the interventionist will perform a brief check in, and may discuss the patient's experience with them for 1-2 minutes after the intervention. Patients will be encouraged to practice the techniques at home between sessions. Patients will also be offered literature on mental health promotion.
  Interventions: Other: Meditation
- Control Group (No Meditation Exposure) (No Intervention): Patients randomized to the control group will be offered literature on mental health promotion and Treatment as Usual in the dialysis setting.

INTERVENTIONS:
Other: Meditation — 10-15 minutes of individually conducted medication practices (silent meditations, guided meditations, body scans, gentle arm movement exercises).
  Arms: Meditation Intervention Arm

SUMMARY:
This study examines the use of brief meditation interventions for patients with symptoms of anxiety and depression who are undergoing dialysis. Half of the participants will receive meditation interventions 3 times a week, while the other half will receive treatment as usual. This study will examine whether meditation is feasible and whether it has any effect on reducing symptoms of anxiety or depression.

DETAILED DESCRIPTION:
Roughly 50% of people who undergo dialysis experience stress, anxiety or depression, but often these conditions go undetected and untreated. It is known that meditation is helpful for anxiety and depression, especially in people who have chronic health conditions. This study will look specifically at meditation interventions tailored to the dialysis setting. Patients on maintenance hemodialysis with anxiety and depression will be recruited from hemodialysis units. Recruitment will start at the Jewish General Hospital in March 2016. Recruitment may later expand to University Health Network (Toronto), and/or other sites affiliated with McGill University or University of Toronto.

Participants will then be randomly assigned to receive meditation or continue with their usual treatment. The participants assigned to the meditation group will practice several meditation techniques with a trained interventionist 3 times a week, during their dialysis sessions.

At the end of the 8 weeks, the investigators will assess whether the meditation intervention was feasible (i.e. whether recruitment goals were met and drop out rates were as expected). Participants in the meditation group will be asked to rate whether they enjoyed the meditation on a scale. Both the participants assigned to the meditation group and to the usual treatment group will be asked to rate their depression and anxiety symptoms on the PHQ-9 and the GAD-7 scales to evaluate whether there was any change.

ELIGIBILITY:
Inclusion Criteria:

* Patients currently receiving maintenance hemodialysis
* Patients with depression and/or anxiety as indicated by scores of ≥10 on the Patient Health Questionnaire (PHQ-9) and/or General Anxiety Disorder-7 (GAD- 7)
* Normal cognition or Mild Cognitive Impairment ("Normal" Result on the 3-minute Mini-Cog Test)

Exclusion Criteria:

* Mild, Moderate, or Severe Dementia ("Abnormal" Result on the 3-minute Mini-Cog Test)
* Acute psychotic symptoms
* Acute Suicidal ideation/intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-03; Primary Completion 2017-12-01 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Proportion of participants screened as eligible who enroll | 34 months
Proportion of participants who enrolled who completed the 8 week-trial | 34 months
Tolerability of Meditation Intervention on a 10-point Likert scale | 8 weeks
  Tolerability of intervention on a 10-point Likert scale

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire (PHQ-9) | Baseline and at 8 weeks
Change in General Anxiety Disorder-7 (GAD-7) | Baseline and at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karl Looper, MD, FRCPC, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Individual data will be coded and anonymized. Anonymized data will not be shared.

REFERENCES:
- [Derived] Natale P, Ju A, Strippoli GF, Craig JC, Saglimbene VM, Unruh ML, Stallone G, Jaure A. Interventions for fatigue in people with kidney failure requiring dialysis. Cochrane Database Syst Rev. 2023 Aug 31;8(8):CD013074. doi: 10.1002/14651858.CD013074.pub2. PMID 37651553